CLINICAL TRIAL: NCT03595930
Title: An Open Label, Multi-centre, Post Marketing Surveillance to Observe the Safety and Effectiveness of ARNUITY Administered in Patients With Asthma in Usual Practice
Brief Title: Post-marketing Surveillance (PMS) Study to Observe the Safety and Effectiveness of ARNUITY in Asthma Subjects in a Real World Setting
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 207435
Record Dates: First submitted 2018-07-12; First posted 2018-07-23 (Actual); Last update posted 2020-08-24 (Actual); Status verified 2020-08

CONDITIONS: Asthma
Keywords: ARNUITY; Effectiveness; Asthma; Post-marketing surveillance; Safety
MeSH Terms: conditions — Asthma | interventions — Fluticasone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 22 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Subjects who received ARNUITY: This PMS will be conducted with subjects who were administered ARNUITY in accordance with the approved label.
  Interventions: Drug: Arnuity

INTERVENTIONS:
Drug: Arnuity — ARNUITY consist of Fluticasone Furoate, is an Inhaled corticosteroids (ICS) medicine taken as one inhalation, once daily, for the control and prevention of asthma in adults and children aged 12 years and older.

SUMMARY:
This is an open-label, multi-center, PMS study to observe the safety and effectiveness of ARNUITY administered in asthma subjects in a real world setting. This PMS shall observe how a broad range of subjects use the drug in the early stages after obtaining the approval. The objective of this PMS is to collect safety and effectiveness data on ARNUITY's approved label in a real world setting. Total of 600 subjects shall be recruited throughout the PMS period; 01 Sep, 2018 to 30 June 2020. ARNUITY is the registered trademark of GSK group of companies.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric subjects older than 12 years of age and adult subjects with asthma
* Subjects who will administer ARNUITY in accordance with the product information approved in Korea
* Subjects who have signed the informed consent form for the PMS

Exclusion Criteria:

* Subjects with status asthmaticus or subjects who have administered ARNUITY as primary therapy for other acute asthmatic episodes that require intensive treatment
* Subjects who have any known hyper-sensitivity to the drug or its ingredients
* Subjects who have severe hypersensitive reactions to milk proteins
* Subjects with hereditary problems of galactose intolerance, the Lapp lactase deficiency, or glucose-galactose malabsorption

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This PMS will be conducted with subjects who were administered ARNUITY in accordance with the approved label. The safety analysis population shall consist of subjects who have administered at least one dose of ARNUITY and have received at least one safety assessment. The effectiveness analysis population shall consist of subjects who have completed the physician's effectiveness assessment (i.e., improved, unchanged, exacerbated, or un-assessable) based on the results of the pulmonary function test or asthma symptom control after administering ARNUITY for 24 weeks (or longer).
Sampling Method: Non-Probability Sample
Enrollment: 668 (Actual)
Dates: Start 2018-09-21 (Actual); Primary Completion 2020-07-22 (Actual); Study Completion 2020-07-22 (Actual)

PRIMARY OUTCOMES:
Incidence rate of adverse events (AEs) after ARNUITY administration | Up to 22months
  An AE is defined as any undesirable, unintended signs (e.g., abnormal laboratory findings), symptoms, or disease that may occur after administration or during use of the product, and does not necessarily have to have a causal relationship with the product.
Incidence rates of unexpected AEs and adverse drug reactions (ADRs) | Up to 22 months
  An ADR is defined as an adverse event whose causal relationship with the product cannot be ruled out.
Incidence rates of serious AEs (SAEs) and serious ADRs (SADRs) | Up to 22 months
  A SAE refers to any one of the following adverse events, which: results in death or is life-threatening; results in or prolongs hospitalization; results in persistent or serious disability or incapacity; results in a birth defect or anomaly; or is an important medical event. SADR is defined a SAE whose causal relationship with the product cannot be ruled out.
Number of subjects with abnormal findings as assessed by physician's effectiveness assessment | Week 24
  For the subjective assessment of effectiveness, the physicians shall assess physician's effectiveness assessment at Week 24 after administration of Arnuity, based on the pulmonary function test and/or asthma symptom control.
Change in Forced Expiratory Volume in 1 Second (FEV1) before and after ARNUITY administration | Week 0, Week 24
  The physicians shall collect FEV1 data at Week 0 and Week 24 after Arnuity administration. The change in the FEV1 results before and after administration of the product shall be analyzed using a paired t-test.
Change in Forced Vital Capacity (FVC) before and after ARNUITY administration | Week 0, Week 24
  The physicians shall collect FVC data at Week 0 and Week 24 after Arnuity administration. The change in the FVC results before and after administration of the product shall be analyzed using a paired t-test.
Change in FEV1/FVC ratio before and after ARNUITY administration | Week 0, Week 24
  The physicians shall collect FEV1/FVC data at Week 0 and Week 24 after Arnuity administration. The change in the FEV1/ FVC ratio before and after administration of the product shall be analyzed using a paired t-test
Changes in the asthma symptom control results before and after ARNUITY administration | Week 0, Week 24
  The physician shall collect the asthma symptom control results at Week 0 and Week 24 after Arnuity administration, based on the symptoms the subjects experienced for the past 4 weeks. The results of the asthma symptom control shall be categorized into 'Controlled', 'Partly Controlled', and 'Uncontrolled'.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com